CLINICAL TRIAL: NCT07315152
Title: Validation of Artificial Intelligence-Driven Cephalometric Analysis as a Reliable Tool for Orthodontic Diagnosis and Treatment Planning
Brief Title: Validation of AI-Based Cephalometric Analysis in Orthodontics
Acronym: AI-CEPH
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hamdi Khalaf Ali, Principal Investigator (Master's Degree Researcher), Al-Azhar University
Other Study IDs: AI-CEPH-VAL-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Malocclusion
Keywords: Treatment planing Orthodontics cephalometric analysis
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients undergoing routine cephalometric analysis, used to validate AI-driven measurements against manual tracings.
  Interventions: Diagnostic Test: Artificial Intelligence-Driven Cephalometric Analysis

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence-Driven Cephalometric Analysis — Cephalometric analysis performed using AI software, compared with manual tracings for validation of accuracy in orthodontic diagnosis and treatment planning.

SUMMARY:
This study is designed to evaluate whether artificial intelligence can analyze cephalometric images in orthodontics as a reliable tool for diagnosis and treatment planning. The study will include orthodontic patients who need cephalometric evaluation. Participants will have their X-ray images analyzed using both the AI system and traditional manual methods. The study will compare the results to see how closely the AI measurements match the standard measurements. This information may help patients, families, and health care providers understand how AI can support orthodontic diagnosis and treatment planning.

DETAILED DESCRIPTION:
Cephalometric analysis is a fundamental diagnostic tool in orthodontics. Conventional manual tracing is time-consuming and operator-dependent, while artificial intelligence-based software has been introduced to improve efficiency and consistency.

This observational study will evaluate and compare manual and AI-assisted cephalometric analyses using lateral cephalometric radiographs. Selected angular and linear measurements will be assessed, and the agreement between the two methods will be statistically analyzed to determine accuracy and reliability.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease.
* Not receiving medical treatment that could interfere with bone metabolism.
* Good level of oral hygiene.
* No periodontal disease or radiographic evidence of bone loss.

Exclusion Criteria:

* Periodontally compromised patients.
* Presence of systemic diseases.
* Drug dependencies.
* Uncooperative patients.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: consists of orthodontic patients aged 12 to 40 years who require orthodontic diagnosis and treatment planning. Participants will have good-quality lateral cephalometric radiographs taken using standardized imaging protocols. The study includes both male and female patients with no previous orthodontic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI-driven cephalometric analysis | Day 1
  Comparison of cephalometric measurements obtained using AI software with manual tracings to evaluate the accuracy and reliability of AI-driven analysis in orthodontic diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Mohammed, DDs,phD, Principal Investigator — Al-Azhar University
Locations (1):
- Faculty of Dentistry, Al-Azhar University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data has not yet been finalized. Considerations regarding participant confidentiality, data protection regulations, and ongoing study procedures may affect the ability to share IPD in the future.

REFERENCES:
- [Background] Kunz F, Stellzig-Eisenhauer A, Zeman F, Boldt J. Artificial intelligence in orthodontics : Evaluation of a fully automated cephalometric analysis using a customized convolutional neural network. J Orofac Orthop. 2020 Jan;81(1):52-68. doi: 10.1007/s00056-019-00203-8. Epub 2019 Dec 18. PMID 31853586
- See also: Scientific and biomedical literature related to orthodontics and artificial intelligence. — https://www.ncbi.nlm.nih.gov